CLINICAL TRIAL: NCT07097571
Title: Comparison of the Efficacy of Proximal and Distal Suprascapular Nerve Blocks Under Ultrasound Guidance in the Treatment of Patients Diagnosed With Adhesive Capsulitis
Brief Title: Suprascapular Nerve Block in the Management of Patients Diagnosed With Adhesive Capsulitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, MUSA AVŞAR, medical doctor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IstanbulUC-MAvsar-01
Record Dates: First submitted 2025-07-25; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Adhesive Capsulitis of the Shoulder; Suprascapular Nerve Block
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients Receiving Suprascapular Nerve Block at the Suprascapular Notch (Active Comparator)
  Interventions: Procedure: Glenohumeral Joint Injection and Suprascapular Nerve Block
- Patients Receiving Suprascapular Nerve Block at the Spinoglenoid Notch (Active Comparator)
  Interventions: Procedure: Glenohumeral Joint Injection and Suprascapular Nerve Block

INTERVENTIONS:
Procedure: Glenohumeral Joint Injection and Suprascapular Nerve Block — An intra-articular injection into the glenohumeral joint will be performed using 4 cc of normal saline and 1 cc of betamethasone. Additionally, a suprascapular nerve block will be administered with 5 cc of lidocaine(%2).

SUMMARY:
This study aims to compare the efficacy of different suprascapular nerve block techniques in patients diagnosed with adhesive capsulitis.

Adhesive capsulitis, commonly known as frozen shoulder, is a condition characterized by pain and restricted range of motion in the shoulder joint, significantly affecting quality of life. The suprascapular nerve provides sensory innervation to the shoulder joint; therefore, nerve blockade is frequently used to alleviate pain. However, there are limited studies evaluating the difference in efficacy between proximal and distal suprascapular nerve blocks.

In this research, two different blockade techniques-at the suprascapular notch and the spinoglenoid notch-will be compared in patients diagnosed with adhesive capsulitis at Istanbul University-Cerrahpaşa between 2024 and 2026. The hypothesis of the study is that the block performed at the spinoglenoid notch provides pain relief comparable to the suprascapular notch block while resulting in less motor blockade.

Patients participating in the study will be randomly assigned to two groups. Both groups will receive an intra-articular corticosteroid injection into the shoulder joint, along with cold application, Codman exercises, and standard medical therapy. Pre- and post-treatment evaluations will include pain severity (NRS), shoulder function (Modified Constant Score), muscle strength, and range of motion.

The results will reveal which technique provides better improvement in shoulder external rotator and abductor muscle strength, shoulder function, and pain relief, thereby offering valuable insights to guide treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had shoulder pain, restricted range of motion (ROM), and night pain for at least 4 weeks

Exclusion Criteria:

* Age younger than 35 years or older than 75 years.
* Known allergy to the agents used for injection.
* History of trauma and/or surgery involving the same shoulder.
* Presence of uncontrolled diabetes mellitus and/or hypertension.
* Presence of severe chronic respiratory disease.
* Presence of severe heart failure.
* Administration of intra- or peri-articular steroid injection to the affected shoulder within the past 2 months.
* Radiographic evidence of calcific tendinitis, glenohumeral osteoarthritis, acromioclavicular joint osteoarthritis, or bone fracture.
* Full-thickness rotator cuff tear detected by shoulder ultrasonography.
* History of surgical intervention or recent/past fracture in the ipsilateral upper extremity.
* Presence of complex regional pain syndrome or vascular disease in the ipsilateral extremity.
* Known coagulation disorders.
* Cervical disc pathology causing radiculopathy.
* Presence of inflammatory or malignant diseases.
* History of cerebrovascular disease.
* Presence of mental impairment or severe psychiatric disorders.
* Pregnancy.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-07-26 (Estimated); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the Strength of Shoulder External Rotation and Abduction. | Patients will be assessed at baseline (pre-procedure), 1 week, and 1 month following the glenohumeral joint injection and suprascapular nerve block
  Shoulder external rotation strength will be assessed in two different positions: with the arm at the side of the body and with the shoulder in 90 degrees of abduction. Additionally, shoulder abduction strength will be evaluated in two positions: with the shoulder in 90 degrees of abduction and in 90 degrees of abduction combined with 30 degrees of horizontal adduction.
Pain Relief | Patients will be evaluated before the glenohumeral joint injection and suprascapular nerve block, as well as 1 hour, 1 week, and 1 month after the procedure.
  Pain will be assessed using the Numerical Rating Scale (NRS), which ranges from 0 (no pain) to 10 (worst pain imaginable), at rest, during movement, at night, and overall, both before and after injections into the glenohumeral joint and suprascapular nerve block. Higher scores indicate worse pain outcomes.
Passive and Active Range of Motion of Shoulder | Patients will be assessed at baseline (pre-procedure), and at 1 hour, 1 week, and 1 month following the glenohumeral joint injection and suprascapular nerve block.
  The shoulder joint's active and passive range of motion will be measured with a goniometer

SECONDARY OUTCOMES:
The Numeric Rating Scale (NRS) | Assessments were performed before, 1 hour after, 1 week after, and 1 month after the glenohumeral joint injection and suprascapular nerve block.
  A pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable
Modified Constant Murley Score | Assessments were performed before, 1 week after, and 1 month after the glenohumeral joint injection and suprascapular nerve block.
  Patients will be assessed according to the modified Constant score, focusing on pain, activities of daily living, range of motion, and muscle strength.
Shoulder Disability Questionnaire | Assessments were performed before, 1 week after, and 1 month after the glenohumeral joint injection and suprascapular nerve block.
  Patients will respond to the items of the Shoulder Disability Questionnaire with reference to the past 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berghs BM, Sole-Molins X, Bunker TD. Arthroscopic release of adhesive capsulitis. J Shoulder Elbow Surg. 2004 Mar-Apr;13(2):180-5. doi: 10.1016/j.jse.2003.12.004. PMID 14997096
- [Background] Wang JP, Huang TF, Hung SC, Ma HL, Wu JG, Chen TH. Comparison of idiopathic, post-trauma and post-surgery frozen shoulder after manipulation under anesthesia. Int Orthop. 2007 Jun;31(3):333-7. doi: 10.1007/s00264-006-0195-7. Epub 2006 Aug 23. PMID 16927088
- [Background] Hamdan TA, Al-Essa KA. Manipulation under anaesthesia for the treatment of frozen shoulder. Int Orthop. 2003;27(2):107-9. doi: 10.1007/s00264-002-0397-6. Epub 2002 Sep 13. PMID 12700935
- [Background] Bae KH, Park KC, Jeong GM, Lim TK. Proximal vs Distal Approach of Ultrasound-guided Suprascapular Nerve Block for Patients With Adhesive Capsulitis of the Shoulder: Prospective Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 May;102(5):819-827. doi: 10.1016/j.apmr.2020.11.003. Epub 2020 Dec 1. PMID 33275962
- [Background] Yildizhan R, Cuce I, Veziroglu E, Calis M. Comparison of Spinoglenoid Versus Suprascapular Notch Approaches for Ultrasound-Guided Distal Suprascapular Nerve Blocks for Shoulder Pain: A Prospective Randomized Trial. Pain Physician. 2024 Jan;27(1):11-19. PMID 38285026
- [Background] Buchbinder R, Green S, Youd JM, Johnston RV, Cumpston M. Arthrographic distension for adhesive capsulitis (frozen shoulder). Cochrane Database Syst Rev. 2008 Jan 23;2008(1):CD007005. doi: 10.1002/14651858.CD007005. PMID 18254123
- [Background] Shanahan EM, Gill TK, Briggs E, Hill CL, Bain G, Morris T. Suprascapular nerve block for the treatment of adhesive capsulitis: a randomised double-blind placebo-controlled trial. RMD Open. 2022 Nov;8(2):e002648. doi: 10.1136/rmdopen-2022-002648. PMID 36418088
- [Background] Jump CM, Waghmare A, Mati W, Malik RA, Charalambous CP. The Impact of Suprascapular Nerve Interventions in Patients with Frozen Shoulder: A Systematic Review and Meta-Analysis. JBJS Rev. 2021 Dec 22;9(12). doi: 10.2106/JBJS.RVW.21.00042. PMID 34936584
- [Background] Zadro J, Rischin A, Johnston RV, Buchbinder R. Image-guided glucocorticoid injection versus injection without image guidance for shoulder pain. Cochrane Database Syst Rev. 2021 Aug 26;8(8):CD009147. doi: 10.1002/14651858.CD009147.pub3. PMID 34435661
- [Background] Lorbach O, Anagnostakos K, Scherf C, Seil R, Kohn D, Pape D. Nonoperative management of adhesive capsulitis of the shoulder: oral cortisone application versus intra-articular cortisone injections. J Shoulder Elbow Surg. 2010 Mar;19(2):172-9. doi: 10.1016/j.jse.2009.06.013. Epub 2009 Oct 1. PMID 19800262
- [Background] Buchbinder R, Hoving JL, Green S, Hall S, Forbes A, Nash P. Short course prednisolone for adhesive capsulitis (frozen shoulder or stiff painful shoulder): a randomised, double blind, placebo controlled trial. Ann Rheum Dis. 2004 Nov;63(11):1460-9. doi: 10.1136/ard.2003.018218. PMID 15479896
- [Background] Buchbinder R, Green S, Youd JM, Johnston RV. Oral steroids for adhesive capsulitis. Cochrane Database Syst Rev. 2006 Oct 18;2006(4):CD006189. doi: 10.1002/14651858.CD006189. PMID 17054278
- [Background] Diercks RL, Stevens M. Gentle thawing of the frozen shoulder: a prospective study of supervised neglect versus intensive physical therapy in seventy-seven patients with frozen shoulder syndrome followed up for two years. J Shoulder Elbow Surg. 2004 Sep-Oct;13(5):499-502. doi: 10.1016/j.jse.2004.03.002. PMID 15383804
- [Background] Page MJ, Green S, Kramer S, Johnston RV, McBain B, Chau M, Buchbinder R. Manual therapy and exercise for adhesive capsulitis (frozen shoulder). Cochrane Database Syst Rev. 2014 Aug 26;2014(8):CD011275. doi: 10.1002/14651858.CD011275. PMID 25157702
- [Background] Ryu KN, Lee SW, Rhee YG, Lim JH. Adhesive capsulitis of the shoulder joint: usefulness of dynamic sonography. J Ultrasound Med. 1993 Aug;12(8):445-9. doi: 10.7863/jum.1993.12.8.445. PMID 8411327
- [Background] Whelton C, Peach CA. Review of diabetic frozen shoulder. Eur J Orthop Surg Traumatol. 2018 Apr;28(3):363-371. doi: 10.1007/s00590-017-2068-8. Epub 2017 Nov 1. PMID 29094212
- [Background] Juel NG, Brox JI, Brunborg C, Holte KB, Berg TJ. Very High Prevalence of Frozen Shoulder in Patients With Type 1 Diabetes of >/=45 Years' Duration: The Dialong Shoulder Study. Arch Phys Med Rehabil. 2017 Aug;98(8):1551-1559. doi: 10.1016/j.apmr.2017.01.020. Epub 2017 Feb 17. PMID 28219686
- [Background] Shaffer B, Tibone JE, Kerlan RK. Frozen shoulder. A long-term follow-up. J Bone Joint Surg Am. 1992 Jun;74(5):738-46. PMID 1624489
- [Background] Hand C, Clipsham K, Rees JL, Carr AJ. Long-term outcome of frozen shoulder. J Shoulder Elbow Surg. 2008 Mar-Apr;17(2):231-6. doi: 10.1016/j.jse.2007.05.009. Epub 2007 Nov 12. PMID 17993282
- [Background] Hazleman BL. The painful stiff shoulder. Rheumatol Phys Med. 1972 Nov;11(8):413-21. doi: 10.1093/rheumatology/11.8.413. No abstract available. PMID 4646489
- [Background] Grey RG. The natural history of "idiopathic" frozen shoulder. J Bone Joint Surg Am. 1978 Jun;60(4):564. No abstract available. PMID 670287
- [Background] Zreik NH, Malik RA, Charalambous CP. Adhesive capsulitis of the shoulder and diabetes: a meta-analysis of prevalence. Muscles Ligaments Tendons J. 2016 May 19;6(1):26-34. doi: 10.11138/mltj/2016.6.1.026. eCollection 2016 Jan-Mar. PMID 27331029
- [Background] Reeves B. The natural history of the frozen shoulder syndrome. Scand J Rheumatol. 1975;4(4):193-6. doi: 10.3109/03009747509165255. PMID 1198072
- [Background] Moren-Hybbinette I, Moritz U, Schersten B. The clinical picture of the painful diabetic shoulder--natural history, social consequences and analysis of concomitant hand syndrome. Acta Med Scand. 1987;221(1):73-82. doi: 10.1111/j.0954-6820.1987.tb01247.x. PMID 2436441